CLINICAL TRIAL: NCT04140032
Title: Addressing Obesity in Early Care and Education Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Roshan Bastani, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-000570
Record Dates: First submitted 2019-10-18; First posted 2019-10-25 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Obesity
Keywords: obesity; nutrition; physical activity; preschool; child care centers; policy-system-environment intervention
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Centers in the group will participate in the A-B-C Healthy Me/Soy Saludable multi- component nutrition and physical activity preschool intervention.
  Interventions: Behavioral: Multi-level preschool obesity control intervention
- Control group (No Intervention): Preschools in the group will continue with "usual care" practices. Control group preschools will receive intervention materials and accompanying instructions after follow-up measures are collected for each cohort.

INTERVENTIONS:
Behavioral: Multi-level preschool obesity control intervention — The multi-level intervention is a preschool-based program that integrates healthy nutrition and physical activity policies and practices into preschool operations via the Sesame Street Healthy Habits for Life curriculum. In addition to the curriculum, the intervention includes coaching sessions to enhance teacher lesson planning to routinely include nutrition and physical activity; as well as assist preschool site directors with implementing policy changes and parent engagement sessions.
  Arms: Intervention group

SUMMARY:
Childhood obesity is a national epidemic that disproportionately burdens low income and ethnic minority populations. By preschool, nearly one-third of low income children are already overweight or obese, setting the stage for adverse health outcomes over their life course. Evidence is mounting that individual-focused, single-component interventions fail to produce long-term population-level changes in obesity-related outcomes. Evidence increasingly supports creating entire environments (e.g., schools) in which the healthy choice is the default option.

The investigators will conduct a pragmatic cluster randomized trial to evaluate the effectiveness of a multilevel (organization, teacher, parent, child) intervention to support healthy eating and physical activity in preschools. The study is being conducted in partnership with Child Care Resource Center (CCRC), a non-profit organization dedicated to ensuring that all children receive high quality preschool experiences. The investigators will randomly assign 60 preschool sites (stratified by size), located in underserved areas of Los Angeles, to the intervention or a usual practice control conditions.

The investigators will evaluate the effectiveness of the intervention on child BMI z-scores (primary outcome) and parent-reported child nutrition and physical activity (secondary outcomes). The investigators will systematically examine the implementation process to understand factors that may facilitate or hinder intervention uptake and success. The findings from this work will be critical for informing future dissemination efforts.

DETAILED DESCRIPTION:
This study involves a 2-group design with stratified cluster randomization at the level of the preschool. The investigators will recruit 60 preschools from LA County's most vulnerable communities, stratified by size (large, small). The investigators will randomly select pairs of schools from each stratum and randomly assign one member of each pair to the intervention or control conditions. Given the 10-month instructional year (Sept. 1-June 30), preschools will be recruited in three cohorts over three instructional years (~20 schools per cohort). To control for time trends in outcomes, the randomization protocol will be implemented independently within each cohort. Baseline data collection, conducted in the first six weeks of the school year, will include surveys (site directors, teachers, parents), anthropometric measures (children), preschool policy reviews and direct observation in preschools including child-level eating behavior and physical activity.

The multilevel intervention will be initiated immediately following baseline data collection and will consist of 1) establishment of organizational policies to support healthy nutrition and physical activity, 2) integration of nutrition and physical activity content into curricula 3) supports for teachers and staff to model healthy behavior, and 4) engagement of parents as partners in implementing healthy policies in preschool and at home. Implementation measures will be collected throughout the project period. Follow-up data collection, in the last four-six weeks of the school year, will mirror baseline data collection.

Study Hypotheses:

1. Children at intervention schools will gain less weight relative to height gains compared to children at control schools, resulting in lower mean BMI z-scores at follow-up (effectiveness). Outcomes will be assessed in the overall sample and among the subset of children who are overweight or obese at baseline.
2. Intervention preschools will have greater implementation of healthy nutrition and physical activity policies and practices at follow-up compared to control preschools.

The primary effectiveness outcome will be child age-and sex-adjusted BMI z-score. The investigators will obtain baseline data on 1,630 children, 815 per condition, 60 preschool site directors and approximately 135 teachers. Estimating 80% child retention at follow-up, the investigators anticipate having follow-up data on 1,304 children, 652 per study arm. Data will also be collected from the parents of participating children at baseline and follow-up.

ELIGIBILITY:
Inclusion Criteria:

Preschool Sites:

* Must be in CCRC network of preschools
* Have 20 or more preschool aged children (2.5-5 years old) in attendance at site
* Children must eat at least one meal on-site per school day
* Must have at least one preschool classroom

Providers (Teachers and Preschool Site Directors):

* Teachers must teach a preschool class at participating preschool
* Be able to provide informed consent

Parents and Children:

* Child must be 2.5-5 years old and enrolled in the participating preschool
* Child primary caregiver must have at least one child 2.5-5 years old that is enrolled in the preschool
* Child primary care giver must be able to read and write in English or Spanish

Exclusion Criteria:

Preschool Sites:

* Have less than 20 preschool aged children (2.5-5 years old) enrolled.
* Do not have a preschool classroom
* Are not in the CCRC network
* Preschools that are based in a family-home or serve special needs children exclusively
* Children do not eat at least one meal on-site per school day

Providers (Teachers and Preschool Site Directors):

-Teachers not currently teaching a preschool class

Parents and Children:

* Child primary care giver unable to read or write in English or Spanish
* Primary care giver who does not have a child currently enrolled in a preschool class

Min Age: 30 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1136 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roshan Bastani, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Fielding School of Public Health, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 68 preschools were screened
Pre-assignment Details: 51 preschools were randomized; 3 withdrew before baseline data collection. All students in a preschool were assigned to the same group.
  The study used an open cohort design in which all students who provided data at baseline and/or follow-up were included. Note: We use the 1136 preschool children included in the primary outcome (BMI z-score)
Units Other Than Participants: Preschool
Groups:
- Intervention: Preschools participated in the A-B-C Healthy Me/Soy Saludable multi-component nutrition and physical activity preschool intervention.
- Control: Preschools continued with "usual care" practices. Control group preschools received intervention materials and accompanying instructions after follow-up measures were collected for each cohort.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 618; 25 Preschool | 518; 23 Preschool
Completed | 618; 25 Preschool | 518; 23 Preschool
Not Completed | 0; 0 Preschool | 0; 0 Preschool

BASELINE CHARACTERISTICS:
Population: All participants for whom valid height, weight, age, and sex were collected at baseline and/or follow-up. The discrepancies between Baseline Participants and results provided in the Baseline Analysis Population Description vary due to missing and/or invalid data presented across demographic categories.
Units Other Than Participants: Preschools
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 601 | 501 | 1102
Number analyzed (Preschools) | 25 | 22 | 47
Age, Customized [Mean (Standard Deviation); unit: Months] — Age measured in months
  Months
    Age, Continuous | 45.3 (9.2) | 43.7 (9.6) | 44.6 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 289 | 224 | 513
  Male | 312 | 277 | 589
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 237 | 195 | 432
  Not Hispanic or Latino | 195 | 178 | 373
  Unknown or Not Reported | 169 | 128 | 297
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 22 | 18 | 40
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 18 | 22 | 40
  White | 96 | 91 | 187
  More than one race | 121 | 94 | 215
  Unknown or Not Reported | 340 | 276 | 616
Region of Enrollment [Number; unit: participants]
  United States | 601 | 501 | 1102

OUTCOME MEASURES:

1. Primary Outcome: Child BMI Z-score
Description: Height and weight of preschool children were measured by trained research staff. These data were used to calculate children's body mass index (BMI) scores.
  The BMI Z-score is a measure calculated from a child's height and weight that indicates how a child's BMI compares with the BMI of a reference population of U.S. children of the same age and sex. The reference population is based on Center for Disease Control and Prevention (CDC) pediatric growth charts and the BMI Z-score is calculated using a CDC-provided computer program. A Z-score of 0 corresponds to the mean BMI of the reference population. A Z-score of +1 corresponds to a BMI that is one standard deviation above the mean of the reference population, and a Z-score of -1 represents a BMI that is one standard deviation below the mean of the reference population. When used as a measure of obesity risk, a lower Z-score is considered a better outcome.
Time Frame: Measured pre-intervention at the beginning of the school year and post-intervention at the end of the school year (approximately 10 months later)
Population: All participants for whom valid height, weight, age, and sex were collected at baseline and/or follow-up.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Intervention | Control
Number analyzed (Participants) | 601 | 501
Z-score
  Baseline | 0.40 (1.07) | 0.43 (1.13)
  Follow-up | 0.31 (1.14) | 0.48 (1.17)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.003, Mixed Models Analysis; p < 0.05 considered significant; Difference between groups in change in B = -0.18, 95% CI 2-sided [-0.31 to -0.06], Standard Deviation 0.06

2. Secondary Outcome: Percentage of Children Who Eat Fruit Once a Day
Description: Parents completed surveys regarding children's physical activity and nutrition. For frequency of fruit consumption, the following question was asked: How often does your child eat... fruit? Include fresh, frozen, or canned fruit. DO NOT include juices. The response is dichotomized as at least once a day versus less than once a day.
Time Frame: as for outcome 1
Population: All participants with a valid response to the survey question at baseline and/or follow-up.
Measure: Number; unit: Percent of children who eat fruits
Arm/Group | Intervention | Control
Number analyzed (Participants) | 425 | 386
Percent of children who eat fruits
  Baseline | 82 | 76
  Follow-up | 86 | 82
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.7, Mixed Models Analysis; p < 0.05 considered significant; Odds ratio for difference between groups = 1.29, 95% CI 2-sided [.034 to 4.91] — Reported dispersion parameter is standard error of log(OR)

3. Secondary Outcome: Frequency of Physical Activity
Description: Parents completed surveys regarding children's physical activity and nutrition. For frequency of physical activity, the following question was asked: During the past 7 days, on how many days was your child physically active for a total of at least 60 minutes per day?
Time Frame: as for outcome 1
Population: All participants with a valid response to the survey question of interest at baseline and/or follow-up.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention | Control
Number analyzed (Participants) | 420 | 379
days
  Baseline | 4.9 (2.1) | 4.8 (2.1)
  Follow-up | 5.2 (2.0) | 5.4 (2.0)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.3, Mixed Models Analysis; Difference between groups in change in f = -0.20, 95% CI 2-sided [-0.58 to 0.17], Standard Deviation 0.19

4. Secondary Outcome: Teacher Nutrition Behaviors
Description: Teacher nutrition will be measured via self-report of dietary intake.
Time Frame: 4 weeks post intervention
Reporting Status: Not Posted

5. Secondary Outcome: Teacher Physical Activity Behaviors
Description: Teacher physical activity will be measured via self-report of physical activity.
Time Frame: 4 weeks post intervention
Reporting Status: Not Posted

6. Secondary Outcome: Nutrition and Physical Activity Policies and Practices at Preschool Site Level
Description: Nutrition and physical activity policies of the preschool will be assessed via in-person all day observations of one preschool classroom per site. Trained research staff will conduct these observations during an on-site visit to the center. Additionally, preschool site directors will complete a nutrition and physical activity policy and practice survey to assess center nutrition and physical activity policies.
Time Frame: 4 weeks post intervention
Reporting Status: Not Posted

7. Secondary Outcome: Percentage of Children Who Eat Vegetables Once a Day
Description: Parents completed surveys regarding children's physical activity and nutrition. For frequency of vegetable consumption, the following question was asked: How often does your child eat... vegetables? DO NOT count potatoes, or beans. The response is dichotomized as at least once a day versus less than once a day.
Time Frame: as for outcome 1
Population: All participants with a valid response to the survey question at baseline and/or follow-up.
Measure: Number; unit: Percentage children who eat vegetables
Arm/Group | Intervention | Control
Number analyzed (Participants) | 424 | 386
Percentage children who eat vegetables
  Baseline | 61 | 61
  Follow-up | 69 | 69
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.8, Mixed Models Analysis; p < 0.05 considered significant; Odds ratio for difference between groups = 1.10, 95% CI 2-sided [0.56 to 2.16], Standard Error of Mean 0.35 — Reported dispersion parameter is standard error of log(OR)
Statistical Analysis 2: Comparison: Intervention vs Control; Test type: Superiority; p = 0.8, Mixed Models Analysis; p < 0.05 considered significant; Odds ratio for difference between groups = 1.10, 95% CI 2-sided [0.56 to 2.16] — Reported dispersion parameter is standard error of log(OR)

ADVERSE EVENTS:
Time Frame: Over the 4 year study period, we recruited 4 cohorts of participants. The period of time over which adverse event data was collected averaged between 8-10 months or the length of the intervention.
Description: This study implemented a multi-level obesity prevention intervention in preschools that posed no risk for serious adverse events or all cause mortality. We monitored for "other" or non-serious adverse events.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/618 | 0/518
Serious Adverse Events (participants affected / at risk) | 0/618 | 0/518
Other Adverse Events (participants affected / at risk) | 0/618 | 0/518

LIMITATIONS AND CAVEATS:
The impact of COVID-19 led to fewer number of participants analyzed in the intervention and control conditions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-12-17): https://cdn.clinicaltrials.gov/large-docs/32/NCT04140032/Prot_000.pdf
  • Statistical Analysis Plan (2025-04-05): https://cdn.clinicaltrials.gov/large-docs/32/NCT04140032/SAP_001.pdf